CLINICAL TRIAL: NCT05069766
Title: Preoperative Marking of the Oral Resection Margin in Esophageal Cancer With a Surgical Fiducial Marker - First Experiences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Nanovi (Unknown)
Responsible Party: Principal Investigator, Trygve Ulvund Solstad, Research Scholar, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-21041919
Record Dates: First submitted 2021-09-15; First posted 2021-10-06 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Esophagus Cancer, Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BioXmark™ (Experimental)
  Interventions: Other: BioXmark™

INTERVENTIONS:
Other: BioXmark™ — During a scheduled outpatient gastroscopy, the tumor margins will be endoscopically marked by BioXmark™. BioXmark™ will be implanted at the most proximal margin of the tumor and 5 cm proximally of the tumor border.

SUMMARY:
This study aims to evaluate if BioXmark™, a surgical marker, may efficiently and safely be used to preoperatively mark the proximal and distal resection line 5 cm proximal and distal to the tumor margin of gastroesophageal-junction adenocarcinoma (GEJ AC).

Furthermore, to determine if placing the resection margin according to the resection margin defined by BioXmark™ is superior to the current standard of a proximal resection line estimation by the individual surgeon based on the intraoperative findings.

DETAILED DESCRIPTION:
In Denmark, the national guidelines for GEJ AC surgery are an R0 resection with a minimum 5 cm proximal and distal resection margin, measured in vivo. During the operation, the primary surgeon sets the resection margin according to the guidelines, with 5 cm on either side.

The Danish national guidelines are clear, but the literature behind them is not, and the recommendations for resection margins vary worldwide. With the lack of a strong literature-backed guideline and a surgical approach that is heavily dependent on the individual surgeon's estimate, the risk of a microscopic positive resection margin (R1 resection) increases. Both problems, namely resectability at the definitive surgery and the incidence of microscopic positive resection margins after resection, may be improved by preoperatively marking the tumor margins in vivo. This could be achieved with an endoscopically placed surgical marker.

One such surgical marker is BioXmark™, a liquid injectable and adherent fiducial marker that has shown promising results for image-guided adaptive radiotherapy in lung, bladder, and esophageal cancer. BioXmark™ is implanted during endoscopy and has appropriate visibility with good positional stability on CT, CBCT, and MRI. Furthermore, no adverse reactions or events have been reported yet.

The study will be performed as a feasibility study of BioXmark™ at the Department of Surgery & Transplantation, Centre of Cancer and Organ Diseases. The investigators plan to include 10 patients who are scheduled to undergo curatively intended surgery for GEJ AC. The patients will be drawn from the existing operating program.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred with gastroesophageal adenocarcinoma to the Department of Surgery & Transplantation, Centre of Cancer and Organ Diseases, Rigshospitalet, and who are candidates for curatively intended surgery.

Exclusion Criteria:

* Patients under the age of 18.
* Patients diagnosed with disseminated disease during surgery.
* Patients with impaired cognitive ability, making obtainment of informed consent impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Registration of visibility of BioXmark™ | From day 0 to the day of operation
  BioXmark™ feasibility in terms of visibility with ultrasound during surgery CT-scans after neoadjuvant and visibility and positional stability during CT-scanning following neoadjuvant chemotherapy preoperatively.
Registration of treatment related side effects assessed by CTCAE V 5.0 | Day 0 to 2 weeks after implantation
  This is part of a safety evaluation and will be registered by CTCAE into Adverse Events (AE) and Serious Adverse Events (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Achiam, MD, DMSCi, Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshopitalet, Department of Surgery and Transplantation, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No